CLINICAL TRIAL: NCT00554801
Title: Central Auditory Processing Disorders Associated With Blast Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C5067-R
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-07

CONDITIONS: Central Auditory Processing Disorder; Traumatic Brain Injury; Hearing Loss
Keywords: Central Auditory Processing; Traumatic Brain Injury; Hearing Loss
MeSH Terms: conditions — Language Development Disorders; Brain Injuries, Traumatic; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blast (Experimental): The study group includes soldiers who have recently been exposed to a high-explosive blast while stationed in Iraq or Afghanistan. They will be recruited at Walter Reed Army Medical Center, Washington, DC. They will undergo audiological testing.
  Interventions: Procedure: Audiological testing
- Control (Active Comparator): Control group are subjects matched to the experimental group by age, gender, and hearing loss, but who have not been exposed to a blast. They will undergo the same audiological testing as the experimental group
  Interventions: Procedure: Audiological testing

INTERVENTIONS:
Procedure: Audiological testing — Subjects will take part in a battery of audiological tests meant to evaluate the function and status of the auditory system. These tests are similar to the kinds of testing carried out routinely in audiology clinics, and include behavioral tests of pure tone hearing, speech perception, and central auditory function, and electrophysiological testing of the middle ear and of the central auditory system.

SUMMARY:
The incidence of central auditory dysfunction in war fighters who are exposed to high-explosive blasts while serving in combat have not been clearly determined. The objectives of this study are to determine whether central auditory processing (CAP) disorders are associated with exposure to high-explosive blasts. This study will also examine the incidence, magnitude and timing of spontaneous recovery of CAP function from blast exposure. The information provided by this study will help guide clinicians in both the military and VA health care systems regarding the likelihood of central auditory processing disorders in soldiers returning from deployment and suggest some clinical rehabilitative strategies for the treatment of these patients with CAP deficits.

DETAILED DESCRIPTION:
The incidence and nature of central auditory dysfunction in combat soldiers who are exposed to high-explosive blasts have not been determined. Using a battery of behavioral and neurophysiological auditory tests, we propose to evaluate central auditory function in soldiers who recently have been exposed to explosive blasts while deployed in Iraq or Afghanistan. In collaboration with the Army Audiology & Speech Center at Walter Reed Army Medical Center (WRAMC), the research will be coordinated at the National Center for Rehabilitative Auditory Research (NCRAR) at the Portland VA Medical Center, and data collection will take place both at the NCRAR and at WRAMC. The study objectives are to determine if specific central auditory processing disorders are often associated with exposure to high-explosive blasts, and if these disorders spontaneously recover or remain over time. One hundred patients who have suffered a blast exposure, but have either no brain damage or mild traumatic brain injury (TBI), will be recruited at WRAMC to participate in this research study. A battery of central auditory processing tests will be administered to participants as soon as possible after their arrival at WRAMC. Patients who demonstrate aspects of central auditory processing disorder will be invited to participate in further testing nine to twelve months later. Those subjects will be brought to the NCRAR at the Portland VA Medical Center or will return to WRAMC for two days of auditory testing, where they will undergo the same battery of tests administered initially. Control subjects who do not have a history of blast exposure and who are matched in age, gender, and audiometric configuration with the experimental subjects will also be tested at the NCRAR site. Data extracted by interview and from medical records, including details of the blast exposure, scores on overall tests of brain function administered by the WRAMC TBI team, presence or absence of post traumatic stress disorder, as well as self-report questionnaires regarding quality of life, presence of tinnitus and/or balance problems, will be used in the interpretation of results.

ELIGIBILITY:
Inclusion Criteria:

Experimental group:

* Active duty soldier at Walter Reed Army Medical Center, Washington DC
* a notation in medical record of exposure to blast
* a Glasgow Coma Scale of 13-15, indicating mild or no traumatic brain injury (TBI
* cognitive and physical ability to take part in these auditory evaluations.
* Age 18 years or older
* native speaker of English (since test materials are presented in English)

Control group:

* able to commute to Portland (Oregon)VA Med Ctr.
* no exposure to blast
* cognitive and physical ability to take part in these auditory evaluations.
* age 18 years or older
* native speaker of English

Exclusion Criteria:

* hearing loss greater than 50 dB HL three-frequency pure tone average bilaterally

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie R. Leek, PhD, Principal Investigator — VA Loma Linda Healthcare System, Loma Linda, CA
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Gallun FJ, Lewis MS, Folmer RL, Diedesch AC, Kubli LR, McDermott DJ, Walden TC, Fausti SA, Lew HL, Leek MR. Implications of blast exposure for central auditory function: a review. J Rehabil Res Dev. 2012;49(7):1059-74. doi: 10.1682/jrrd.2010.09.0166. PMID 23341279
- [Result] Gallun FJ, Diedesch AC, Kubli LR, Walden TC, Folmer RL, Lewis MS, McDermott DJ, Fausti SA, Leek MR. Performance on tests of central auditory processing by individuals exposed to high-intensity blasts. J Rehabil Res Dev. 2012;49(7):1005-25. doi: 10.1682/jrrd.2012.03.0038. PMID 23341276
- See also: Web site of the American Speech-Language Hearing Association — http://www.asha.org
- See also: web site of Defense and Veterans Brain Injury Center — http://www.dvbic.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Active duty military who were exposed to a blast while deployed and were patients at Walter Reed Army Medical Center; only mild or no traumatic brain injury
Groups:
- Blast-exposed: The study group includes soldiers who have recently been exposed to a high-explosive blast while stationed in Iraq or Afghanistan. They will be recruited at Walter Reed Army Medical Center, Washington, DC.
  Audiological testing: Subjects will take part in a battery of audiological tests meant to evaluate the function and status of the auditory system. These tests are similar to the kinds of testing carried out routinely in audiology clinics, and include behavioral tests of pure tone hearing, speech perception, and central auditory function, and electrophysiological testing of the middle ear and of the central auditory system.
- Control Group: No exposure to high-intensity blast; matched to blast-exposed group on gender, age, and hearing loss
Period: Overall Study
Arm/Group | Blast-exposed | Control Group
Started | 55 | 29
Completed | 36 | 29
Not Completed | 19 | 0
Not completed — left area before completion | 5 | 0
Not completed — Withdrawal by Subject | 14 | 0

BASELINE CHARACTERISTICS:
Population: All participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Blast-exposed | Control Group | Total
Number analyzed (Participants) | 36 | 29 | 65
Age, Continuous [Mean (Full Range); unit: years] | 32.8 [20 to 54] | 32.1 [19 to 54] | 32.5 [19 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 32 | 26 | 58
Region of Enrollment [Number; unit: participants]
  United States | 36 | 29 | 65

OUTCOME MEASURES:

1. Primary Outcome: Audiological Test Results
Description: Audiometric testing, with normal hearing specified as better (lower) than 25 decibels Hearing Level (dBHL), and a mild hearing loss between 25 to 50 dBHL.
Time Frame: three years
Measure: Mean (Standard Deviation); unit: decibels Hearing Level
Arm/Group | Blast-exposed | Control Group
Number analyzed (Participants) | 36 | 29
decibels Hearing Level | 10.8 (6.0) | 6.6 (4.2)

2. Secondary Outcome: Quality of Life Questionnaire
Description: Self-report questionnaires regarding quality of life
Time Frame: Three years
Population: It was decided early during implementation of this study that the investigators would not collect self-report data on quality of life, so there are no data to report
Groups:
- Blast-exposed: Soldiers who have been exposed to one or more blasts
- Controls: Individuals who have not experienced a blast
Arm/Group | Blast-exposed | Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Blast-exposed | Control Group
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/29
Other Adverse Events (participants affected / at risk) | 0/55 | 0/29

LIMITATIONS AND CAVEATS:
A quality-of-life self-report questionnaire was not implemented for this study, and so no data on this outcome were collected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes